CLINICAL TRIAL: NCT04691375
Title: A Phase 1a/1b Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PY314 as a Single Agent and In Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: A Study of PY314 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor business decision.
Sponsor: Ikena Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PY314-1-01
Record Dates: First submitted 2020-12-08; First posted 2020-12-31 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor; Gynecologic Cancer; Breast Cancer; Colorectal Cancer; Lung Adenocarcinoma; Renal Cell Carcinoma; Triple Negative Breast Cancer; Hormone Receptor/Growth Factor Receptor-Negative Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Adenocarcinoma of Lung; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Ovarian Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Part A: Dose escalation of PY314 alone and in combination with pembrolizumab in a standard 3+3 design
  Part B: Dose expansion of one or more dose levels of PY314 administered alone and in combination with pembrolizumab for predefined tumor histology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part A: PY314 Single agent dose level 1 (Experimental): PY314 single agent dose level will depend on any safety signal observed in this cohorts only. Following the determination of the safety and tolerability of at least two PY314 dose levels by the safety review committee.
  Interventions: Drug: PY314
- Part A: PY314 Single agent dose level 2 (Experimental): PY314 single agent dose level 2 dose escalation of PY314 as a single agent will continue in the absence of unacceptable dose limiting toxicity to the maximum administered dose as defined in the predefined dose escalation schema.
  Interventions: Drug: PY314
- Part A: PY314 Single agent dose level 3 (Experimental): PY314 single agent dose level 3 to identify the maximum tolerated dose and/or to determine the recommended dose for expansion of PY314
  Interventions: Drug: PY314
- Part A: PY314 Single agent dose level 4 (Experimental): PY314 single agent dose level 4 to characterize the pharmacokinetic profile of PY314 as a single agent.
  Interventions: Drug: PY314
- Part A: Combination dose level 1 (Experimental): Combination dose level 1 to characterize the safety and tolerability of PY314 as a single agent and in combination with pembrolizumab in subjects with advanced refractory solid tumors including refractory to check point inhibitor.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part A: Combination dose level 2 (Experimental): PY314 combination dose level 2 to identify the maximum tolerated dose and/or to determine the recommended dose for expansion of PY314 administered alone and in combination with pembrolizumab.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part A: Combination dose level 3 (Experimental): PY314 combination dose level 3 to characterize the pharmacokinetic profile of PY314 as a single agent and in combination with pembrolizumab.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part A: Combination dose level 4 (Experimental): PY314 combination dose level 4 to describe, in subjects selected by pre-specified tumor histology, anti-tumor activity of PY314 administered alone and in combination with pembrolizumab.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part B: Single agent dose expansion dose level 1 (Experimental): PY314 single agent dose expansion dose level 1 to define further the safety and tolerability of PY314 alone.
  Interventions: Drug: PY314
- Part B: Combination dose expansion cohort 1 (Experimental): PY314 in combination with pembrolizumab dose expansion cohort 1 to define the safety and tolerability of PY314 alone and in combination with pembrolizumab over multiple treatment cycles in subjects with pre-defined tumor histologies and confirmed TREM2 expression.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part B: Combination dose expansion cohort 2 (Experimental): PY314 in combination with pembrolizumab dose expansion cohort 2 to further characterize the PK profile of PY314 as a single agent and in combination with pembrolizumab.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part B: Combination dose expansion cohort 3 (Experimental): PY314 in combination with pembrolizumab dose expansion cohort 3 to characterize the anti-tumor activity of PY314 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM2 expression.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part B: Combination dose expansion cohort 4 (Experimental): PY314 in combination with pembrolizumab dose expansion cohort 4 to evaluate the incidence of ADA formation and TREM2 expression.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab
- Part B: Combination dose expansion cohort 5 (Experimental): PY314 in combination with pembrolizumab dose expansion cohort 5 to further explore and characterize the anti-tumor activity of PY314 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM2 expression.
  Interventions: Drug: Combination Therapy: PY314 + Pembrolizumab

INTERVENTIONS:
Drug: PY314 — Dose of PY314 as a single agent given in a standard 3+3 design.
  Arms: Part A: PY314 Single agent dose level 1; Part A: PY314 Single agent dose level 2; Part A: PY314 Single agent dose level 3; Part A: PY314 Single agent dose level 4; Part B: Single agent dose expansion dose level 1
Drug: Combination Therapy: PY314 + Pembrolizumab — Dose of PY314 alone and given in combination with pembrolizumab
  Other Names: PY314; Pembrolizumab
  Arms: Part A: Combination dose level 1; Part A: Combination dose level 2; Part A: Combination dose level 3; Part A: Combination dose level 4; Part B: Combination dose expansion cohort 1; Part B: Combination dose expansion cohort 2; Part B: Combination dose expansion cohort 3; Part B: Combination dose expansion cohort 4; Part B: Combination dose expansion cohort 5

SUMMARY:
This is an open-label, multicenter, first in human, Phase 1a/1b study of PY314 in subjects with locally advanced (unresectable) and/or metastatic solid tumors that are refractory or relapsed to standard of care (including pembrolizumab, if approved for that indication).

DETAILED DESCRIPTION:
Part A: Dose escalation of PY314 alone and in combination with pembrolizumab in a standard 3+3 design Part B: Dose expansion of one or more dose levels of PY314 administered alone and in combination with pembrolizumab for predefined tumor histology

ELIGIBILITY:
KEY ELIGIBILITY CRITERIA

Inclusion Criteria:

* Adults ≥18 years of age at the time of study consent
* Subjects with any of the following eligible solid tumor diagnoses as confirmed by cytology or histology:

  * Escalation Cohorts (Part A): Subjects with advanced solid tumors from pre-specified tumor types (Gynecological cancers [including ovarian, fallopian, primary peritoneal, endometrial, cervical, vaginal, vulvar], gastric [adenocarcinoma], Colorectal ([MSIlow and CPI refractory MSIhigh]), lung [non-small cell lung adenocarcinoma and squamous cell carcinoma] who are recurrent or refractory to platinum-based chemotherapy in addition to prior treatment with CPI Programmed Cell Death-1 (PD-1)/Programmed Cell Death-Ligand 1 (PD-L1) or who give informed consent to forego such therapy, renal [clear cell and non-clear cell], breast [TNBC and HR+ HER-2-] with locally advanced or metastatic disease that is relapsed or refractory to at least one line of post-adjuvant therapy (including a CPI-either alone or in combination if approved for that indication, and not eligible for other targeted therapies specific for their tumor type).
  * Expansion Cohorts (Part B): Subjects with advanced solid tumors selected from 5 prespecified cancers based on preclinical and Part A.
* Subjects must provide an original, diagnostic tumor sample to determine TREM2 expression (sites have verified source prior to screening and availability of archival tissue during screening). Subjects without an archival tissue sample will only be eligible if they choose and consent to provide a CNB of primary or a metastatic lesion required for part B, used in Part A only if an archival specimen unavailable.
* Subjects must have documented disease progression (including prior treatment with a CPI (alone or in combination), if approved for that indication.
* There is no limit to the number of prior treatments.
* Measurable disease by RECIST 1.1
* All acute toxic effects of any prior antitumor therapy, including immunotherapy, have resolved to Grade < 2 before the start of study drug dosing (including Grade < 2 alopecia or peripheral neuropathy, or if controlled on thyroid replacement therapy).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
* Coagulation: International Normalized Ratio (INR) ≤ 1.3, unless on a therapeutic anticoagulant
* Adequate hematologic function defined as follows: Platelets ≥ 100 x 10^9/L; Hemoglobin ≥ 8.0 g/dL; ANC ≥ 1.5 x 10^9/L (without granulocytic growth factors within the previous 7 days of obtaining the screening hematologic laboratory values)
* Adequate hepatic function defined as follows: AST / ALT ≤ 2.5 x upper limit of normal (ULN) (if liver metastases are present, ≤ 5 x ULN); Total or conjugated bilirubin ≤ 1.5 x ULN
* Adequate renal function defined as follows: Serum Creatinine ≤ 2 x ULN or creatinine clearance (CrCl) ≥45 mL/min as calculated by the Cockroft-Gault method

Exclusion Criteria:

* Subject is a candidate for molecularly targeted therapy (e.g., drugs targeting EGFR, VEGF, ALK, ROS-1, NTRK, MET, RET and BRAF V600E, HER2). Applies to enrolled subjects on both Part A and Part B of the study.
* History of autoimmune disorder requiring ongoing or intermittent disease-modifying therapy excluding thyroid disease otherwise well controlled on replacement therapy
* Stable treated or asymptomatic brain metastases for at least 3 months documented by brain imaging prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, active SARS-CoV-2 infection, active or chronic bleeding event within 28 days prior to first dose of study drug, or psychiatric illness/social situation that would limit compliance with study requirements as judged by treating physician
* Decompensated liver disease as evidenced by hepatic encephalopathy or coagulopathy
* Active angina or Class III or IV CHF (NYHA CHF Functional Classification System) or clinically significant cardiac disease within 12 months of first dose of study drug, including MI, unstable angina, Grade 2 or greater peripheral vascular disease, CHF, uncontrolled HTN, or arrhythmias not controlled by medication
* Any anti-cancer therapy, including small molecules, immunotherapy, chemotherapy, monoclonal antibody therapy (except for bone-modifying agents as supportive care), radiotherapy, or any other agents to treat cancer within 21 days (dependent upon the agent and drug half-life), of first dose of study drug
* Refractory lung cancer subjects who have progressed within 3 months of initiating chemotherapy-doublet regimens or lung cancer subjects who have progressed within 6 months of initiation immunotherapy-chemotherapy combination treatment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) | 36 months
  Adverse Events will be summarized by MedDRA system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment related AEs, Serious Adverse Events (SAEs), discontinuations due to AEs, and AEs of at least NCI CTCAE grade 3 severity.
(Part A only) Dose Limiting Toxicity of PY314 | Assessed during first 21 days of treatment
  Evaluation of dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Measure PY314 concentration at the end of infusion (CEOI) | 36 months
  Measure PY314 concentration at the end of infusion (CEOI) after the first dose.
Measure PY314 concentration at the trough level (Ctrough) | 36 months
  Measure PY314 concentration at the trough level (Ctrough). All subjects who received at least 1 dose of PY314 and have at least 1 measured concentration at a scheduled PK time point after start of dosing.
Determining PY314 time to maximum concentration (Tmax) | 36 months
  Determining PY314 time to maximum concentration (Tmax) during Cycle 1.
Measure PY314 Area under the curve (AUC)0-t | 36 months
  Measure PY314 Area under the curve (AUC)0-t. All subjects who received at least 1 dose of PY314 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Measure PY314 half-life (T1/2) | 36 months
  Measure PY314 half-life (T1/2). All subjects who received at least 1 dose of PY314 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Measure PY314 Clearance (CL) | 36 months
  Measure PY314 Clearance (CL). All subjects who received at least 1 dose of PY314 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Measure PY314 Volume at Steady State (Vss) | 36 months
  Measure PY314 Volume at Steady State (Vss). All subjects who received at least 1 dose of PY314 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Measure PY314 maximum concentration (Cmax) | 36 months
  Measure PY314 maximum concentration (Cmax) at various time points during Cycle 1. All subjects who received at least 1 dose of PY314 and have at least 1 measured concentration at a scheduled PK time point after start of dosing.
Incidence of Anti-Drug Antibody (ADA) formation to PY314 | 36 months
  To evaluate the incidence of anti-drug antibody (ADA) formation to PY314
Objective response rate (ORR) | 36 months
  The incidents of ORR is defined as either a complete or partial response per RECIST. Subjects with no baseline data will be considered no responders. ORR will be summarized by dose, tumor type, and overall. ORR will be summarized descriptively.
Clinical Benefit Rate (CBR) | 36 Months
  Defined as the percentage of subjects who have achieved complete response, partial response and stable disease.
Duration of response (DOR) | 36 months
  DOR will be calculated to determine durability. DOR will be measured from the time by which the criteria for CR or PR-whichever is recorded first-are met until the first date by which recurrent or progressive disease is objectively documented. DOR will be assessed using KAPLAN-MEIER methods.

OTHER OUTCOMES:
Progress free survival (PFS) | 36 months
  PFS will be measure from entry onto the study until disease progression or death from any cause. PFS will be assessed using KAPLAN-MEIER methods.
Overall survival (OS) | 36 months
  The duration of overall survival (OS) will be measured from the time of first study drug administration until the date of death. OS will be assessed using KAPLAN-MEIER methods.

CONTACTS AND LOCATIONS:
Overall Officials: Len Reyno, MD, Study Director — Ikena Oncology; Marc Chamberlain, MD, Study Director — Ikena Oncology
Locations (23):
- United States (23):
  - Mayo Clinic Scottsdale - PPDS, Phoenix, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope - Comprehensive Cancer Center, Duarte, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - OHSU Knight Cancer Institute Beaverton Clinic, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Start South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Wisconsin Institutes for Medical Research, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beckermann KE, Patnaik A, Winer I, Tan W, Bashir B, Kyriakopoulos CE, Sweis RF, Chamberlain M, Rini BI. A phase 1b open-label study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of py314 in combination with pembrolizumab in patients with advanced renal cell carcinoma. Invest New Drugs. 2024 Apr;42(2):179-184. doi: 10.1007/s10637-024-01419-1. Epub 2024 Feb 19. PMID 38372949
- [Derived] Binnewies M, Pollack JL, Rudolph J, Dash S, Abushawish M, Lee T, Jahchan NS, Canaday P, Lu E, Norng M, Mankikar S, Liu VM, Du X, Chen A, Mehta R, Palmer R, Juric V, Liang L, Baker KP, Reyno L, Krummel MF, Streuli M, Sriram V. Targeting TREM2 on tumor-associated macrophages enhances immunotherapy. Cell Rep. 2021 Oct 19;37(3):109844. doi: 10.1016/j.celrep.2021.109844. PMID 34686340